CLINICAL TRIAL: NCT01862250
Title: Phase I-II Clinical Trial to Determine the Safety of Clonidine in Infants With Hypoxic Ischemic Encephalopathy During Therapeutic Hypothermia
Brief Title: Safety of Clonidine in Infants With Hypoxic Ischemic Encephalopathy During Therapeutic Hypothermia
Acronym: HIE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID: NA_00072308; NCT02252848 (obsolete NCT alias)
Record Dates: First submitted 2013-04-01; First posted 2013-05-24 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Encephalopathy, Hypoxic-Ischemic
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Clonidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clonidine infants with HIE (Experimental): Infants in this group will receive Intravenous clonidine at 1µg/kg/dose either every 6 or 8 hrs from the start of cooling to the end of re-warming
  Interventions: Drug: Clonidine (Duraclon®)

INTERVENTIONS:
Drug: Clonidine (Duraclon®) — Clonidine at dosing intervals of 6, 8, 12, 18 or 24 hours. If the following is observed the event will be recorded, and no additional clonidine will be given and blood will be drawn to measure plasma level of clondine.
  * 10 mm Hg reduction in MAP or MAP ≤ 40 mm Hg sustained for ≥30 min after administration
  * 20% drop in HR from the infant's baseline, sustained for ≥30 min after administration
  * HR ≤70/min, sustained for ≥30 min after administration

SUMMARY:
This research is being done to find out the safety of the investigational study drug, Clonidine Hydrochloride ( CLON). , in infants who are undergoing whole body cooling for the treatment of hypoxic ischemic encephalopathy (HIE). The only known and effective treatment for HIE is therapeutic hypothermia or whole body cooling for72 hours. During the cooling process, babies get agitated, shiver and are uncomfortable. To treat these side effects morphine is frequently used. CLON is very effective in decreasing shivering in adults and children. Furthermore, in some preclinical studies, clonidine has been shown to be neuroprotective (safe for the brain in models of brain injury)..This is a Phase I-II to determine if low dose CLON will reduce the incidence of shivering and whether it has short term cardiovascular safety. In this Phase I-II study, the investigators will determine the (i) the maximum tolerated dose of CLON during cooling for HIE, (ii) the effects of CLON on heart rate, blood pressure, core body temperature and cerebral autoregulation (ability to maintain constant blood flow to the brain) and (iii) association between blood levels and changes in the above parameters. In this study the investigators hope to find ways to improve sedation, shivering and agitation in newborn infants with HIE on the cooling protocol. Our ultimate goal is determine the potential neuro-protective properties of clonidine in newborn babies with HIE.

DETAILED DESCRIPTION:
The most desirable sedative-analgesic agent used in infants with HIE would 1) have an excellent safety profile, 2) provide adequate analgesia and sedation, 3) reduce shivering, 4) cause minimal respiratory depression, 5) preserve cerebrovascular autoregulation, and 6) confer neuroprotection. Several lines of evidence suggest alpha 2 adrenergic receptor agonist class of sedatives-analgesics may have all these properties. The investigators have recently developed a sensitive assay to measure clonidine levels which will allow us to perform population Pharmacokinetic (PK)/Pharmacodynamic (PD) analyses of clonidine in sick newborns. Thus, this phase I/II trial is designed to test the hypothesis clonidine , an alpha- 2 adrenergic receptor agonist, will reduce the incidence of shivering without adversely affecting heart rate (HR), blood pressure (BP), temperature regulation or cerebrovascular autoregulation.

Essentially all classes of sedative-analgesic agents affect mean arterial blood pressure (MAP) which can alter cerebral perfusion and affect cerebrovascular autoregulation. Cerebrovascular autoregulation is when blood flow to the brain is held relatively constant over a wide range of MAPs; it ensures a steady supply of oxygenated blood to the brain, and is only functional within a specific range of MAP's. When MAP deviates from this range and drops below the lower limit of autoregulation, blood flow becomes passive to MAP and the brain is placed at risk for ischemic injury. Brain injury alters cerebrovascular autoregulation in the region of injury, and together with sub-optimal MAP after hypoxic brain injury could cause more brain ischemia leading to poor outcomes, seizures, and permanent neurologic injuries. Little information is available on the effect of HIE alone or in combination with hypothermia on cerebrovascular autoregulation, and no information is published on the direct effect of sedative-analgesics on alterations in hemodynamic parameters and subsequent indirect or direct effects on cerebrovascular autoregulation in newborns with HIE. Thus, this study will establish the safety of clonidine, a commonly used sedative-analgesic in infants and children, in a population of infants with HIE undergoing therapeutic hypothermia. A secondary exploratory outcome is to determine the efficacy of clonidine in reducing shivering during the cooling phase of the therapeutic hypothermia protocol.

ELIGIBILITY:
Inclusion Criteria:

* Infants ≥35 0/7 weeks gestation with the diagnosis of HIE who are being treated with therapeutic hypothermia, who have indwelling arterial lines
* Informed parental consent

Exclusion Criteria:

* Infants who are considered moribund and the clinical team is considering withdrawal of support
* Infants who need > 20 µg/kg/min of dopamine or the addition of epinephrine or dobutamine to maintain a mean arterial pressure (MAP) ≥ 45 mmHg, or milrinone for cardiovascular support
* Baseline heart rate (HR) <80 bpm during hypothermia
* Infants suspected of major chromosomal anomalies, except trisomy 21
* Infants with major cardiovascular anomalies
* Infants with severe persistent pulmonary hypertension of the newborn who are enrolled and who then need Extracorporal Membrane Oxygenation (ECMO) will be withdrawn from the study

Ages: 35 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2013-10-03 (Actual); Primary Completion 2015-04-14 (Actual); Study Completion 2015-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Estelle B Gauda, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agthe AG, Kim GR, Mathias KB, Hendrix CW, Chavez-Valdez R, Jansson L, Lewis TR, Yaster M, Gauda EB. Clonidine as an adjunct therapy to opioids for neonatal abstinence syndrome: a randomized, controlled trial. Pediatrics. 2009 May;123(5):e849-56. doi: 10.1542/peds.2008-0978. Epub 2009 Apr 27. PMID 19398463
- [Background] Angeles DM, Wycliffe N, Michelson D, Holshouser BA, Deming DD, Pearce WJ, Sowers LC, Ashwal S. Use of opioids in asphyxiated term neonates: effects on neuroimaging and clinical outcome. Pediatr Res. 2005 Jun;57(6):873-8. doi: 10.1203/01.PDR.0000157676.45088.8C. Epub 2005 Mar 17. PMID 15774841
- [Background] Roka A, Melinda KT, Vasarhelyi B, Machay T, Azzopardi D, Szabo M. Elevated morphine concentrations in neonates treated with morphine and prolonged hypothermia for hypoxic ischemic encephalopathy. Pediatrics. 2008 Apr;121(4):e844-9. doi: 10.1542/peds.2007-1987. PMID 18381513
- [Background] Zhang Y. Clonidine preconditioning decreases infarct size and improves neurological outcome from transient forebrain ischemia in the rat. Neuroscience. 2004;125(3):625-31. doi: 10.1016/j.neuroscience.2004.02.011. PMID 15099676
- [Background] Shankaran S, Laptook AR, Ehrenkranz RA, Tyson JE, McDonald SA, Donovan EF, Fanaroff AA, Poole WK, Wright LL, Higgins RD, Finer NN, Carlo WA, Duara S, Oh W, Cotten CM, Stevenson DK, Stoll BJ, Lemons JA, Guillet R, Jobe AH; National Institute of Child Health and Human Development Neonatal Research Network. Whole-body hypothermia for neonates with hypoxic-ischemic encephalopathy. N Engl J Med. 2005 Oct 13;353(15):1574-84. doi: 10.1056/NEJMcps050929. PMID 16221780

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study medication was not administered for one participant
Groups:
- Clonidine Infants With HIE: Infants in this group will receive Intravenous clonidine at 1µg/kg/dose either every 6 or 8 hrs from the start of cooling to the end of re-warming
  Clonidine (Duraclon®): Clonidine at dosing intervals of 6, 8, 12, 18 or 24 hours.
  If the following is observed the event will be recorded, and no additional clonidine will be given and blood will be drawn to measure plasma level of clondine.
  * 10 mm Hg reduction in Mean Arterial Pressure (MAP) or MAP ≤ 40 mm Hg sustained for ≥30 min after administration
  * 20% drop in Heart Rate (HR) from the infant's baseline, sustained for ≥30 min after administration
  * HR ≤70/min, sustained for ≥30 min after administration
Period: Overall Study
Arm/Group | Clonidine Infants With HIE
Started | 12
Completed | 8
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Groups:
- Clonidine Infants With HIE: Infants in this group will receive Intravenous clonidine at 1µg/kg/dose either every 6 or 8 hrs from the start of cooling to the end of re-warming
  Clonidine (Duraclon®): Clonidine at dosing intervals of 4, 6, 8, 12, 18 or 24 hours.
  If the following is observed the event will be recorded, and no additional clonidine will be given and blood will be drawn to measure plasma level of clondine.
  * 10 mm Hg reduction in MAP or MAP ≤ 40 mm Hg sustained for ≥30 min after administration
  * 20% drop in HR from the infant's baseline, sustained for ≥30 min after administration
  * HR ≤70/min, sustained for ≥30 min after administration
Arm/Group | Clonidine Infants With HIE
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: weeks] | 38.2 [35.9 to 39.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Steady State Clonidine Blood Levels During Hypothermia
Description: Trough clonidine blood levels were measured after 4-7 doses of clonidine were given intravenously with a dosing interval of every 8 hrs. Mean and standard deviation (SD) of the number of doses given prior to levels being drawn was 5.3 (mean) and 0.37 (SD).
  Time after last dose before measurement was 9hrs (mean) and 2.7hrs (SD).
Time Frame: 3 days
Population: Only 8 babies were assessed for this outcome because the rest did not have a steady state trough level performed during cooling
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Clonidine Infants With HIE
Number analyzed (Participants) | 8
ng/ml | 0.6 [0.27 to 1.06]

2. Primary Outcome: Amount of Morphine Given
Description: Intravenous morphine (mg/kg) was given. The standard dose is 0.05 mg/kg per dose
Time Frame: Up to 2 days
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Clonidine Infants With HIE
Number analyzed (Participants) | 8
mg/kg | 0.02 [0.00 to 0.08]

3. Secondary Outcome: Presence of Shivering After Clonidine
Description: Babies were assessed after administration of clonidine for the presence or absence of shivering.
Time Frame: 48hrs
Measure: Count of Participants; unit: Participants
Arm/Group | Clonidine Infants With HIE
Number analyzed (Participants) | 12
Participants | 0

4. Secondary Outcome: Time to Passive Rewarming
Description: Following 2 hours of therapeutic hypothermia, the temperature of the thermo-blanket is adjusted up half degree per hour allowing passive rewarming until 36.5 degrees is reached
Time Frame: Beginning at 72 hours up to 12 hours
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Clonidine Infants With HIE
Number analyzed (Participants) | 8
Hours | 8.7 [7.4 to 10.1]

ADVERSE EVENTS:
Arm/Group | Clonidine Infants With HIE
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes